CLINICAL TRIAL: NCT02736110
Title: Registry of Celution Device for the Processing of Adipose Derived Regenerative Cells (ADRCs) for Intra-articular Delivery to Knees With Osteoarthritis
Brief Title: Registry of Celution Device for the Processing of Adipose Derived Regenerative Cells (ADRCs) to Treat Osteoarthritis
Acronym: RELIEVE
Status: Withdrawn | Type: Observational
Why Stopped: Corporate decision
Sponsor: Cytori Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: RELIEVE
Record Dates: First submitted 2016-03-15; First posted 2016-04-13 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, knee
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
This registry study will compile information from patients that are scheduled to receive or have received Adipose Derived Regenerative Cells (ADRCs) prepared by the Celution device to treat osteoarthritis in the knee.

ELIGIBILITY:
Inclusion Criteria:

* Males or females > 18 years of age
* Diagnosis of osteoarthritis in one or both knees with Kellgren Lawrence grade ≥ 2 at x-ray evaluation or MRI findings of degenerative changes
* Pain with or without swelling in the affected area for >4 months

Exclusion Criteria:

* Know spine or disc disease or symptomatic nerve impingement contributing to pain in the affected limb
* History of documented nerve damage in the affected limb
* Pregnant or lactating status. Pregnancy as determined by a positive pregnancy test prior to procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are schedule to receive or have received Adipose Derived Regenerative Cells (ADRCs) prepared by the Celution device to treat osteoarthritis in the knee.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change in knee pain as assessed by the knee injury and osteoarthritis outcome score (KOOS) | 90 days

SECONDARY OUTCOMES:
Change in knee pain as assessed by the knee injury and osteoarthritis outcome score (KOOS) | Days 7, 30, 180 and 365
Change in knee pain assessed by VAS Assessments | Days 7, 30, 90, 180 and 365
Change in knee function as assessed by the Lysholm Knee Scoring Scale | Days 7, 30, 90, 180 and 365
Change in WORMS scoring (Whole Organ MRI of the knee) | Days 180 and 365
Change in knee function as measured by Tegner Activity Scale | Days 7, 30, 90, 180 and 365
Change in knee function as measured by the Lower Extremity Functional Scale | Days 7, 30, 90, 180 and 365

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kesten, Study Chair — Cytori Therapeutics

IPD SHARING:
Plan to Share IPD: Yes